CLINICAL TRIAL: NCT03131713
Title: Impact of Preoperative Acetaminophen and Carbohydrate Loading to on Pain and Functional Status in Patients Undergoing Mohs Micrographic Surgery for Non-melanoma Skin Cancers
Brief Title: Preoperative Acetaminophen and Carbohydrate Loading
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12136
Record Dates: First submitted 2017-03-06; First posted 2017-04-27 (Actual); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Non-melanoma Skin Cancer
Keywords: Mohs micrographic surgery; pain; functional status
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will receive usual perioperative care including patient education on diagnosis, treatment and prognosis of skin cancer, encouragement of food and fluid intake prior to and during the surgery as needed, and acetaminophen per patient request.
- Intervention (Experimental): The intervention group, in addition to usual care, will receive Acetaminophen 1000mg and commercially available carbohydrate drink (two pouches of Gatorade Prime Sports Fuel drink containing 50gm carbohydrate in approximately 250ml fluid total) at the beginning of the surgery.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen 1000mg
  Arms: Intervention

SUMMARY:
The study's goal is to assess impact of preoperative acetaminophen and oral carbohydrate drinks on pain and functional status experienced by patients undergoing Mohs micrographic surgery for non-melanoma skin cancers. Patients are randomly assigned to receive standard of care or preoperative acetaminophen 1000 mg and Gatorade sports drinks 2 packets before surgery. Patients are then asked to rate their level of pain, anxiety, thirst, hunger, fatigue on a scale of 0-100 on day of surgery before surgery has started, after clearance of skin cancer, and at the end of the visit. Patients are contacted by phone 48 hours after their surgery to assess their maximum level of post-operative pain (rated from 0-100), usage of over the counter or prescribed pain medications, and presence of complications e.g. bleeding, infection, dehiscence. Differences in perioperative functional status and pain medication usage are compared between patients in control and intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing Mohs micrographic surgery for non-melanoma skin cancers (basal cell carcinoma and squamous cell carcinoma)

Exclusion Criteria:

* history of liver transplant, hepatitis, or cirrhosis, those required to be NPO for subsequent closure by other surgical specialties, or those with known allergy to acetaminophen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bichchau Nguyen, M.D., Principal Investigator — Tufts Medical Center/Tufts University School of Medicine
Locations (1):
- Tufts Dermatology, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events during pre-assignment stage
Period: Overall Study
Arm/Group | Control | Intervention
Started | 50 | 51 (1 intervention subject was added on after the protocol was initiated.)
Completed | 45 | 51
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 45 | 51 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 51 | 96
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (12) | 65 (10) | 65 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 27 | 37 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 45 | 51 | 96
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 51 | 96
Pain scale [Mean (Standard Deviation); unit: units on a pain scale] — Rated on a pain scale of 0-100. Higher score means worse outcome; lower score means better outcome.
  units on a pain scale | 3.4 (1.5) | 1.3 (0.6) | 1.7 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Pain Score
Description: Rated on a pain scale of 0-100. Higher score means worse outcome; lower score means better outcome.
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: units on a pain scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 45 | 51
units on a pain scale | 2.8 (1.1) | 1.2 (0.6)

2. Secondary Outcome: Thirst
Description: Rated on a thirst scale of 0-100. Higher score means worse outcome; lower score means better outcome.
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: score on a thirst scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 45 | 51
score on a thirst scale | 9.4 (18.7) | 10.5 (20.5)

3. Secondary Outcome: Hunger
Description: Rated on a hunger scale of 0-100. Higher score means worse outcome; lower score means better outcome.
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: units on a hunger scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 45 | 51
units on a hunger scale | 19.9 (29.3) | 17.9 (28.3)

4. Secondary Outcome: Anxiety
Description: Rated on n anxiety scale of 0-100. Higher score means worse outcome; lower score means better outcome.
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: score on an anxiety scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 45 | 51
score on an anxiety scale | 7.6 (16.7) | 2.2 (8.3)

5. Secondary Outcome: Fatigue
Description: Rated on a fatigue scale of 0-100. Higher score means worse outcome; lower score means better outcome.
Time Frame: Day of surgery
Measure: Mean (Standard Deviation); unit: score on a fatigue scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 45 | 51
score on a fatigue scale | 12 (18) | 10.7 (18.4)

6. Secondary Outcome: Number of Participants Using Post-operative Analgesic
Description: Number of participants using over the counter and prescribed non-opioid and opioid pain medications
Time Frame: 48 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 45 | 51
Participants | 27 | 34

7. Secondary Outcome: Maximum Post-op Pain Score
Description: Rated on a maximum post-op pain scale of 0-100. Higher score means worse outcome; lower score means better outcome.
Time Frame: 48 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a maximum post-op scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 45 | 51
score on a maximum post-op scale | 14 (22.2) | 13.6 (20)

ADVERSE EVENTS:
Time Frame: 1 year
Description: All-Cause Mortality was not monitored/assessed.
Groups:
- Control; Intervention: The intervention group, in addition to usual care, will receive Acetaminophen 1000mg and commercially available carbohydrate drink (two pouches of Gatorade Prime Sports Fuel drink containing 50gm carbohydrate in approximately 250ml fluid total) at the beginning of the surgery.
  Acetaminophen: Acetaminophen 1000mg
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/51
Other Adverse Events (participants affected / at risk) | 0/45 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT03131713/Prot_SAP_000.pdf